CLINICAL TRIAL: NCT02046564
Title: A Multicenter, Randomized, Double-blind Trial to Assess the Efficacy and Safety of ASC-01 in Patients With Major Depressive Disorder
Brief Title: Assess the Efficacy and Safety of ASC-01 in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-12-005; JapicCTI-142413 (Other: Japic)
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASC-01 (Experimental): The dose of 3-12mg/100mg(Aripiprazole/Sertraline Combination)will be orally administered once daily
  Interventions: Drug: ASC-01
- Placebo (Placebo Comparator): The dose of 0mg/100mg (Placebo/Sertraline Combination ）will be orally administered once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC-01
  Arms: ASC-01
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and the safety of ASC-01 (aripiprazole/sertraline combination) compared to sertraline monotherapy in patients with major depressive disorders who have responded incompletely to sertraline monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are either inpatients or outpatients.
* Patients who are able to understand necessary information for giving consent to undergo examinations, observations, and evaluations specified in this clinical protocol, and who are able to give written consent based on a full understanding of the trial.
* Patients who have been given a diagnosis of "Major Depressive Disorder, Single Episode" or "Major Depressive Disorder, Recurrent" according to the DSM-5 and who have a current episode of major depression that has been continuing for at least 8 weeks
* Patients with a HAM-D 17 total score of 18 or more at the Screening Period evaluation

Exclusion Criteria:

* Female patients of childbearing potential who wish to become pregnant during the trial period or within 4 weeks after completion or discontinuation of the trial
* Pregnant or breast-feeding female patients, or female patients who may be pregnant
* Patients judged to be intolerant to all antidepressant (including drugs not used for their current episodes of major depression) based on their treatment history
* Patients who have had electroconvulsive therapy
* Patients who have enrolled in a clinical trial of other drugs or medical devices within 1 month before the time of informed consent
* Patients who have a medical history suggesting a risk of developing serious adverse events or symptoms that may hinder efficacy/safety evaluation (eg, symptoms of fibromyalgia, or premenstrual syndrome etc that overlap with depressive symptoms)
* Patients with complications or a history of diabetes mellitus, or patients who have been judged to be diabetic

  * fasting blood glucose level ≥ 126 mg/dL
  * 2-hour glucose level in 75-g oral glucose tolerance test (OGTT) ≥ 200 mg/dL
  * non-fasting blood glucose level ≥ 200 mg/dL
  * HbA1c [NGSP level] ≥ 6.5%
* Patients who are undergoing treatment for thyroid disease (except for patients whose disease has been stabilized with drug therapy for 3 months or longer before the time of informed consent)
* Patients who have a history of neuroleptic malignant syndrome or serotonin syndrome
* Patients who have a history of seizure disorder (eg, epilepsy)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 412 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (29):
- Australia (2):
  - Everton Park, Queensland
  - Melbourne
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region
- Malaysia (4):
  - Ipoh
  - Johor Bahru
  - Kuala Lumpur
  - Kuching
- South Korea (9):
  - Busan
  - Chungcheongnam-do
  - Deagu
  - Gangwon-do
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Jeollabuk-do
  - Seoul
- Taiwan (7):
  - Chiayi City
  - Kaohsiung City
  - Keelung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

RESULTS

PARTICIPANT FLOW:
Groups:
- ASC-01: * Formulation A: ASC-01 (aripiprazole/sertraline combination) 3 mg/100 mg tablet
  * Formulation B: ASC-01 (aripiprazole/sertraline combination) 6 mg/100 mg tablet
  * Formulation C: ASC-01 (aripiprazole/sertraline combination) 9 mg/100 mg tablet
  * Formulation D: ASC-01 (aripiprazole/sertraline combination) 12 mg/100 mg tablet Formulation A or, B, C, or D was orally administered once daily. For Week 1, Formulation A was administered after which administration was conducted according to the dose-increase criteria. The formulation was fixed from Week 5 to Week 6.
Period: Overall Study
Arm/Group | ASC-01 | Placebo
Started | 209 | 203
Completed | 194 | 183
Not Completed | 15 | 20
Not completed — Adverse Event | 6 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Subject met withdrawal criteria | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASC-01 | Placebo | Total
Number analyzed (Participants) | 208 | 203 | 411
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 208 | 203 | 411
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.8) | 39.5 (11.8) | 38.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 72 | 151
  Male | 129 | 131 | 260
Region of Enrollment [Number; unit: participants]
  South Korea | 36 | 42 | 78
  Japan | 157 | 142 | 299
  Taiwan | 7 | 10 | 17
  Malaysia | 6 | 5 | 11
  Australia | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated scale which evaluates the level of depression. The MADRS consists of 10 items assessing apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thought. Each item is scored from 0 to 6, with higher scores indicating worse condition.Summed subscales are combined to compute a total score. Total score ranges from 0 to 60, with higher score indicating worse condition.
Time Frame: 8 weeks after the start of the sertraline treatment period (Baseline), 6 weeks after the start of the double-blind period (Last Observation Carried Forward [LOCF])
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
units on a scale | -9.2 (0.5) | -7.2 (0.5)

2. Secondary Outcome: The Montgomery-Åsberg Depression Rating Scale (MADRS) Response Rate
Description: The MADRS is a clinician-rated scale which evaluates the level of depression. The MADRS consists of 10 items assessing apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thought. Each item is scored from 0 to 6, with higher scores indicating worse condition.
  MADRS Response Rate is the percentage of subjects who achieved a decrease in the MADRS total score by 50% or more.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
percentage of participants | 37.5 | 25.6

3. Secondary Outcome: The Montgomery-Åsberg Depression Rating Scale (MADRS) Remission Rate
Description: The MADRS is a clinician-rated scale which evaluates the level of depression. The MADRS consists of 10 items assessing apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thought. Each item is scored from 0 to 6, with higher scores indicating worse condition.
  MADRS Remission Rate is the percentage of subjects who achieved a decrease in the MADRS total score by 50% or more and whose MADRS total score is 10 points or less.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
percentage of participants | 29.3 | 20.2

4. Secondary Outcome: The Clinical Global Impression - Improvement (CGI-I) Improvement Rate
Description: The CGI-I Scale is a clinician-rated scale which assesses the total improvement of the patient's condition compared to that at baseline. Scores range from 0 to 7: 0 = Not assessed, 1= Very much improved, 2 = Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse. Higher scores indicate worse condition. CGI-I Improvement Rate is the percentage of subjects whose CGI-I score is 1 or 2.
Time Frame: 6 weeks after the start of the double-blind period (Last Observation Carried Forward [LOCF])
Measure: Number; unit: percentage of participants
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
percentage of participants | 46.2 | 34.5

5. Secondary Outcome: The Mean Change From Baseline in the Clinical Global Impression - Severity of Illness (CGI-S)
Description: The CGI-S Scale is a clinician-rated scale which assesses how mentally ill the patient is at the time. Scores range from 0 to 7: 0 = Not assessed, 1= Normal, not at all ill, 2 =Borderline mentally ill, 3= Mildly ill, 4= Moderately ill, 5= Markedly ill, 6= Severely ill, 7= Among the most extremely ill patients. Higher scores indicate worse condition.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
units on a scale | -1.0 (0.1) | -0.8 (0.1)

6. Secondary Outcome: The Mean Change From Baseline in the Hamilton Depression Rating Scale 17 (HAM-D17) Total Score
Description: The HAM-D is a clinician-rated scale which evaluates the level of depression. The HAM-D consists of 17 items such as depression mood, feeling of guilt, suicide, insomnia, work and activities, retardation, and so on.
  Each item is scored from 0 to 2, 3 or 4, with higher scores indicating worse condition. Summed subscales are combined to compute a total score. Total score ranges from 0 to 52, with higher score indicating worse condition.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
units on a scale | -6.8 (0.4) | -5.6 (0.4)

7. Secondary Outcome: The Mean Change From Baseline in the Social Adaptation Self-evaluation Scale (SASS) Total Score
Description: The SASS is a self-rating scale which assesses the social motivation and behavior in participants with depression. The SASS consists of 21 items covering the different aspects of social interactions, global social attitude, and self-perception. Each item is scored from 0 to 3, with higher scores indicating better condition.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 164 | 149
units on a scale | 3.7 (0.3) | 1.5 (0.3)

8. Secondary Outcome: The Mean Change From Baseline in the Apathy Scale (AS) Total Score
Description: The AS consists of 14 items. Items 1-8 are scored as follows: 3= Not at all, 2= Slightly, 1= Some, 0= A lot. Items 9-14 are scored as follows: 0= Not at all, 1= Slightly, 2= Some, 3= A lot. Total score ranges from 0-42, with higher score indicating worse condition.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 164 | 149
units on a scale | -3.3 (0.4) | -1.1 (0.4)

9. Secondary Outcome: The Mean Change From Baseline in the Self-rating Version of Montgomery-Åsberg Depression Rating Scale (MADRS-S) Total Score
Description: The MADRS-S is a patient-reported scale based on MADRS, administered to evaluate the level of depression. This scale consists of 9 items assessing patients' mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life. Each item is scored from 0 to 3, with higher scores indicating worse condition. Summed subscales are combined to compute a total score. Total score ranges from 0 to 27, with higher score indicating worse condition.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ASC-01 | Placebo
Number analyzed (Participants) | 208 | 203
units on a scale | -2.85 (0.22) | -1.86 (0.23)

ADVERSE EVENTS:
Time Frame: Double-blind period (6 weeks)
Arm/Group | ASC-01 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/203
Serious Adverse Events (participants affected / at risk) | 0/209 | 2/203
Other Adverse Events (participants affected / at risk) | 128/209 | 107/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASC-01 (N=209) | Placebo (N=203)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASC-01 (N=209) | Placebo (N=203)
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 9 | 10
Stomatitis (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3
Drug withdrawal syndrome (General disorders) | 5 | 3
Nasopharyngitis (Infections and infestations) | 28 | 23
Alanine aminotransferase increased (Investigations) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 1
Weight increased (Investigations) | 9 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 5
Akathisia (Nervous system disorders) | 27 | 7
Dizziness (Nervous system disorders) | 10 | 10
Headache (Nervous system disorders) | 8 | 13
Somnolence (Nervous system disorders) | 5 | 5
Tremor (Nervous system disorders) | 12 | 11
Insomnia (Psychiatric disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No